CLINICAL TRIAL: NCT04009928
Title: Deep Brain Stimulation of the Medial Forebrain Bundle and Subcallosal Cingulate for the Treatment of Treatment Resistant Depression
Brief Title: Deep Brain Stimulation for Treatment Resistant Depression
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Surgeon-Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 277-2018
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: After 6 months of open-label stimulation, patients will enter a blinded, randomized, crossover phase. After a 1 week washout phase with stimulation turned OFF, patients will randomly be assigned to receive 2 weeks of sham stimulation followed by 2 weeks of active stimulation (at their optimized settings), or vice versa.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent researcher will perform the randomization and institute the sham/active stimulation, allowing for continued blinding of participants/care providers/investigators/outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active followed by sham stimulation (Experimental): 2 weeks of active stimulation of the medial forebrain bundle or subcallosal cingulate at the optimized stimulation settings derived during the open-label phase. After 1 week of washout period (with no stimulation), subjects undergo 2 weeks of sham stimulation
  Interventions: Device: Active stimulation of the medial forebrain bundle or subcallosal cingulate; Device: Sham stimulation
- Sham followed by active stimulation (Sham Comparator): 2 weeks of sham-stimulation, followed by 2 weeks of active stimulation, separated with 1 week washout period.
  This is a crossover study, patients will undergo both arms, the order of which they do is randomized.
  Interventions: Device: Active stimulation of the medial forebrain bundle or subcallosal cingulate; Device: Sham stimulation

INTERVENTIONS:
Device: Active stimulation of the medial forebrain bundle or subcallosal cingulate — Deep brain stimulation of the medial forebrain bundle or subcallosal cingulate
Device: Sham stimulation — Sham stimulation for 2 weeks (Cross-over design)

SUMMARY:
Treatment resistant depression (TRD) is a major global health concern, and there is a crucial need to develop novel effective treatments.

The medial forebrain bundle (MFB) is a recently described DBS target, with reported rapid onset of antidepressant effects. A recent small randomized trial reported a 100% response rate. The subcallosal cingulate cortex (SCC) is the most commonly used target in DBS for depression.

Herein, the investigators will conduct a sham-controlled randomized trial of DBS to the MFB or SCC for TRD.

DETAILED DESCRIPTION:
Eight patients with TRD will be treated with DBS to the MFB. At approximately 2 weeks postoperartively, stimulation will be initiated in all patients. Voltage and contact position will be altered initially, looking for optimal and stabilized responses in depressive symptoms, while trying to minimize any side effects.

Following this 6 month open-label optimization phase, patients will be then undergo randomization to receive 2 weeks of stimulation followed by 2 weeks of sham stimulation, or vice versa. These 2 week phases will be separated by a 1 week washout period. Depressive symptoms will be evaluated at the end of each 2 week phase, then patients will resume open-label stimiulation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥20 and ≤80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study Psychiatrist and the surgeon.
3. DSM-V diagnosis of major depressive disorder or bipolar II,
4. At least 5-year illness history of the primary disorder and at least 6 months since the onset of the first episode of major depression.
5. A minimum score of 20 on the Hamilton Depression Rating Scale (HAMD) when depressed)
6. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by two psychiatrists associated with the study. Including specifically:

   1. Failed to respond or tolerate adequate trial of three or more medications accepted as first line in the treatment of depression
   2. Failed to respond or tolerate augmentation with or combination of at least 2 medications known to be first line treatments for depression
   3. An adequate trial of cognitive behavioural therapy or other evidence-supported psychotherapy, delivered by a therapist experienced in treating depression
7. A consistent dose of any and all medications in the 30 days prior to study entry.
8. Women of childbearing potential must agree to use a contraception method throughout the study.

Exclusion Criteria:

1. Past or current evidence of psychosis or mania
2. Active neurologic disease, such as epilepsy
3. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
4. Current active suicidal ideation
5. Any contraindication to MRI scanning
6. Presence of significant cognitive impairment
7. Likely to relocate or move out of the country during the study's duration
8. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure.
9. Currently pregnant (as determined by history and serum HCG) or lactating; for females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Safety: Qualitative report of any adverse events occurring up until 6 months postoperatively | 6 months
  Report of all adverse events (minor and major), including perioperative, followup, and stimulation-related
Proportion of responders as measured by the Hamilton Depression Score (17-item version) at 6 months | 6 months
  Proportion of patients who have a 40% or greater reduction in their Hamilton Depression Score at 6 months compared to their preoperative baseline score.
  The Hamilton Depression score is a 17-item score ranging from 0-50, with lower numbers being less severe.

SECONDARY OUTCOMES:
Mean Hamilton Depression Score (17-item version) at the end of the sham-stimulation compared with at the end of the true-stimulation | 6 months
  At 6 months there is a blinded crossover portion of the study. The Hamilton depressions score will be measured at the end of each of the arms. The score after each arm will be compared.
  The Hamilton Depression score is a 17-item score ranging from 0-50, with lower numbers being less severe.
Hamilton Depression score (17-item version) at 12 months | 12 months
  Proportion of patients with 40% or greater decrease in Hamilton Depression Score at 12 months compared to baseline. The Hamilton Depression score is a 17-item score ranging from 0-50, with lower numbers being less severe.
Montgomery Asberg Depression Depression Rating Scale at 12 months | 12 months
  Proportion of patients with 40% or greater reduction in their Montgomery Asberg Depression Depression Rating Scale at 12 months compared to preoperative baseline. This scale is a 10-item scale with total scores ranging from 0-60, higher numbers being more severe.
Beck Depression Inventory at 12 months | 12 months
  Mean Beck Depression Inventory at 12 months compared to mean beck depression inventory at baseline. The Beck Depression Inventory is a 21-item scale with total scores ranging from 0-63, with lower numbers being more severe than higher.
Short Form (36) Health Survey (SF-36) at 12 months | 12 months
  Comparing mean SF-36 score at 12 months to baseline. The Short-form health survey (36) is a 36-item survey, which produces a total score which is normalized to a score of 0-100 (mean 50), with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada